CLINICAL TRIAL: NCT06850311
Title: Efficacy and Safety of Herbal Topical Ointment in Treating Atopic Dermatitis: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Herbal Ointment in Treating Atopic Dermatitis Topically
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: En Chu Kong Hospital (Other)
Responsible Party: Principal Investigator, Chi-Wen Huang, MD, attending physician of department of Traditional Chinese medicine, En Chu Kong Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ECKIRB1130403
Record Dates: First submitted 2025-02-23; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Atopic Dermatitis; Atopic Dermatitis (AD); Atopic Dermatitis (Eczema); Atopic Dermatitis Eczema; TCM; Skin Diseases; Skin Diseases, Eczematous; Skin Diseases, Genetic
MeSH Terms: conditions — Dermatitis, Atopic; Eczema; Skin Diseases; Skin Diseases, Eczematous; Skin Diseases, Genetic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- herbal ointment (Experimental): 1. Form: ointment
  2. Dose: each gram of ointment contains TCM
  3. Dosing schedule: apply 0.5g of ointment per 10 x 10 dermatitis lesion twice daily
  Interventions: Drug: herbal ointment; Drug: Placebo
- placebo ointment (Placebo Comparator): 1. Form: ointment
  2. Dose: vehicle
  3. Dosing schedule: apply 0.5g of ointment per 10 x 10 dermatitis lesion twice daily
  Interventions: Drug: herbal ointment; Drug: Placebo

INTERVENTIONS:
Drug: herbal ointment — Every 10 x 10 cm area of lesion requires 0.5 g of ointment, applied twice daily (morning and evening, separated by approximately 12±2 hours) for 4 weeks
Drug: Placebo — Every 10 x 10 cm area of lesion requires 0.5 g of ointment, applied twice daily (morning and evening, separated by approximately 12±2 hours) for 4 weeks.

SUMMARY:
Atopic dermatitis (AD), also known as atopic eczema, is a chronic inflammatory skin disorder. The current first-line recommended treatment for AD is the use of emollients, topical corticosteroids (TCS), and oral antihistamines if necessary. However, patients often have side effects like skin atrophy and telangiectasia. And there were plenty of herbal medicine which are beneficial to atopic dermatitis in ancient Chinese medicine books and records. Therefore, the purpose of this study is to develop a new topical application of traditional Chinese medicine and evaluate its clinical efficacy in AD patients. In human trial, 66 Subjects diagnosed as AD will be enrolled and treated with Sophora flavescens Aiton topical ointment. After treatment we will estimate the efficacy and record adverse events to conduct statistically analysis.

The 1st year project: (1) Expect to enroll 66 clinical subjects of AD. (2) Evaluate subjects 'symptom and proceed herbal ointment treatment. (3) Record treatment responses including adverse effect. (4) Conduct statistically analysis.

The 2nd year project: (1) Completing enrollment of 66 clinical subjects of AD. (2) Finish evaluation and treatment of all subjects. (3) Statistically analysis all collecting data (4) Discuss and analyze the outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18 and 65 years old, female or male.
2. Atopic dermatitis fulfilling the diagnostic criteria of Hanifin&Rajka.
3. Atopic dermatitis involving <10% of BSA. (Base on the BSA result of Screening)
4. An Investigator's Global Assessment (IGA) score of 2, 3 or 4 which corresponds to mild, moderate or severe disease. (Base on the IGA result of Screening)
5. Female patients of child-bearing age with negative pregnancy test at screening.
6. Female patients of child-bearing age that agree to continue using birth control measures approved by the investigator and agree not to lactate for the duration of the study.

Agree to only receive stable doses of an additive-free, basic bland emollient for at least 7 days before baseline (day0) Willing to comply with study protocol and agree to sign an informed consent form.

Exclusion Criteria:

1. Having a history of topical or systematical hypersensitivity to herbal or its excipient (e.g. vehicle) in ointment
2. Undergoing phototherapy (e.g. UVB, PUVA) or systemic therapy (e.g. Immunosuppressive agents) within 30 days.
3. Having used topical or oral therapy (e.g. topical corticosteroids, antibiotic, TCM) for dermatitis within 7 days before the first application of the study medication.
4. Having a significant concurrent disease, such as: significant abnormalities in hematology, severe uncontrolled metabolic syndrome (e.g., hypertension, diabetes mellitus, metabolic arthritis, hyperthyroidism), psychiatric disease, cancer or AIDS.
5. Having abnormal liver or renal function (AST/ALT >3 x ULN, creatinine >2.0 mg/dl).
6. Women who are lactating, pregnant or preparing to be pregnant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Percentage change in Eczema Area Severity Index (EASI) scores from baseline to week 4 | 4 weeks
  The Eczema Area and Severity Index (EASI) is used to measure the disease severity of erythema, infiltration/papulation, excoriation, and lichenification each on a scale of 0 to 3 (none to severe) as well as the percentage of disease area on a scale of 0 to 6 for the head ⁄ neck, upper limb, trunk and lower limb body regions. Each body region score is calculated by multiplying the disease severity score by the disease area score and by the multiplier. The scores are summed to give the total EASI score, ranging from 0 to a maximum 72. The mean percentage change in EASI = (EASI baseline-EASI post-treat) / EASI baseline x 100%

SECONDARY OUTCOMES:
Proportion of subjects who have achieved EASI-50, EASI-75, and EASI-90 after 4 weeks of treatment | 4 weeks
  It is defined as at least 50%, 75%, and 90% reduction in EASI score relative to the baseline.
The mean change in Dermatology Life Quality Index (DLQI)from baseline to week 4 | 4 weeks
  The DLQI is a self-administered 10-item questionnaire, ranges from 0 (best) to 30 (worst); the higher the score, the more quality of life is impaired.
Visual Analogue Scale (VAS) for pruritus severity rates | 4 weeks
  from 0 (no itching) to 10 (very severe itching)
The mean percentage change in Total Body Surface Area involved with AD (BSA, range 0%-100%) from baseline to week 4 | 4 weeks
  BSA is total Body Surface Area involved, ranging from 0% (none) to 100% (total body surface involved)
Proportion of subjects with a change in Investigator's Global Assessment (IGA, range 0-5 from baseline to week 4. ) | 4 weeks
  1. Proportion of subjects with an IGA score of 0 (clear) or 1 (almost clear) at week 6.
  2. Proportion of subjects with ≥ 2 point improvement in IGA at week 4.
TCMBCQ (Time Frame: Change from Baseline TCMBCQ at 4weeks) | 4 weeks
  Traditional Chinese Medicine Body Constitution Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- En Chu Kong hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
primary and secondary outcome of this study
Supporting Information: ICF, CSR
Time Frame: information sharing after paper published
Access Criteria: all in public, without any kind of review